CLINICAL TRIAL: NCT03357887
Title: Prognostic Value of Three New Biomarkers of Multiple Sclerosis Compared to Reference Biomarker in Patients With Radiologically Isolated Syndrome
Brief Title: Prognostic Value of Three New Biomarkers of Multiple Sclerosis in Patients With Radiologically Isolated Syndrome
Acronym: T-RIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016/ET-01
Record Dates: First submitted 2017-11-14; First posted 2017-11-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis; Radiologically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of cerebrospinal fluid and serum — Analysis of biomarkers in patient biological samples

SUMMARY:
To look at the prognostic value of new biomarkers in CSF and serum for characterisation of multiple sclerosis

ELIGIBILITY:
Inclusion criteria

* Patients have given their free consent for use of their samples in research
* Patients have at least 2 years of clinical and radiological follow-up data available Exclusion criterion
* No follow-up of patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from whom prospective samples have been collected and conserved in the biobank at Nice as part of the RISC (Radiologically Isolated Syndrome Consortium).
  100 patients with Radiologically Isolated Syndrome as diagnosed by MRI using the Okuda 2009 criteria (65 RIS-: not converted after at least 2 years of follow-up; 35 RIS+).
  30 patients with recurrent-remittent multiple sclerosis 30 symptomatic control patients 20 control patients with inflammatory disease 20 control patients with non-inflammatory neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Level of tumour necrosis factor receptor in cerebrospinal fluid | Baseline
  ELISA
Level of Neurofilament in cerebrospinal fluid | Baseline
  ELISA
Level of GFAP in cerebrospinal fluid | Baseline
  ELISA
Level of secreted glycoprotein in cerebrospinal fluid | Baseline
  ELISA

SECONDARY OUTCOMES:
Level of tumour necrosis factor receptor in serum | Baseline
  ELISA
Level of Neurofilament in serum | Baseline
  ELISA
Level of GFAP in serum | Baseline
  ELISA
Level of secreted glycoprotein in serum | Baseline
  ELISA
Comparison of the conversion time according to the threshold value of each biomarker for Radiologically Isolated Syndrome patients | Baseline
  Log-rank test
Compare prognostic value of all four markers of the high risk criteria (age below 37, male, myelitis). | Baseline
  Multivariate analysis
Biomarker levels in CSF and serum in different patient subpopulations (Radiologically Isolated Syndrome, recurrent remittent MS, symptomatic controls, central nervous system inflammatory disease controls, non-inflammatory disease controls) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Thouvenot E, Hinsinger G, Demattei C, Uygunoglu U, Castelnovo G, Pittion-Vouyovitch S, Okuda D, Kantarci O, Pelletier D, Lehmann S, Marin P, Siva A, Lebrun C. Cerebrospinal fluid chitinase-3-like protein 1 level is not an independent predictive factor for the risk of clinical conversion in radiologically isolated syndrome. Mult Scler. 2019 Apr;25(5):669-677. doi: 10.1177/1352458518767043. Epub 2018 Mar 22. PMID 29564952